CLINICAL TRIAL: NCT06487299
Title: Iron Administration Via Colonic Transendoscopic Enteral Tubing Combined With Washed Microbiota Transplantation for Iron Deficiency:A Double-blind Randomized Controlled Trial
Brief Title: Iron Administration Via Colonic TET Combined With WMT for ID
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TET- RCT-Fe
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Iron Deficiency Anemia in Childbirth
Keywords: Iron; Transendoscopic enteral tubing; Washed Microbiota Transplantation; iron deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous lactate; Ferric Oxide, Saccharated; Saline Solution; Sodium Chloride; Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ferrous Lactate (Experimental): Ferrous lactate is administered via the colon as an injectable solution at a dose of 300 mg per day for 3 days, with saline added to 50ml.
  Interventions: Drug: Ferrous Lactate
- Iron Sucrose (Active Comparator): Iron sucrose is administered via the colon as an injectable solution at a dose of 300mg per day for 3 days, with saline added to 50ml.
  Interventions: Drug: Iron sucrose
- Saline (Placebo Comparator): 0.9% sodium chloride is administered via the colon as an injectable solution at a dose of 50ml per day for 3 days.
  Interventions: Drug: 0.9% NaCl solution

INTERVENTIONS:
Drug: Ferrous Lactate — The injection solution was 3 ferrous lactate (10ml:0.1g iron) mixed with 20ml saline.
  Other Names: PURAMEX(R)
  Arms: Ferrous Lactate
Drug: Iron sucrose — The injection was 3 shots of ferrous lactate (5ml:100mg iron) mixed with 35ml saline.
  Other Names: Iron saccharate
  Arms: Iron Sucrose
Drug: 0.9% NaCl solution — The same volume and color as Iron sucrose.
  Other Names: saline (medicine)
  Arms: Saline

SUMMARY:
The colon can absorb iron.We propose an integrated approach utilizing colonic transendoscopic enteral tubing to deliver iron in different valence states, coupled with washed microbiota transplantation . This clinical trial aims to assess the feasibility, safety, and efficacy of this approach for the treatment of iron deficiency.

DETAILED DESCRIPTION:
At least 60 subjects who meet all the inclusion criteria but do not meet any exclusion criteria will be enrolled in this study. Data of demographic characteristics, reticulocyte hemoglobin, ferritin and clinical outcomes will be collected. After treatment, they will enter the follow-up period for safety and efficacy evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. ferritin ≤30 μg/L;
2. feasible colonic TET placement (cephalic end in the ileocecal region);
3. completion of 3 WMT sessions.

Exclusion Criteria:

1. The patient has other co-morbidities that can lead to iron deficiency, such as acute gastrointestinal haemorrhage and menorrhagia.etc.
2. People who are allergic to iron or taking oral medications that interfere with iron absorption.
3. Patients with heart, brain, lung, liver, kidney and other serious diseases;
4. Patients do not cooperate to complete the clinical trial process;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-07-25 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Reticulocyte haemoglobin values in blood | Baseline; Day 4
  To compare the level of reticulocyte haemoglobin in the blood before and after administration of iron lactate, iron sucrose and saline.

SECONDARY OUTCOMES:
Serum ferritin levels | Baseline; Day 4
  To compare the level of ferritin in the serum before and after administration of iron lactate, iron sucrose and saline.

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline; Day 4
  The number of adverse reactions that are associated with iron medicine reported by subjects from the start of treatment to the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Faming, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Department of Microbiota Medicine & Medical Centre for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Lu AD, Zhang LP, Zuo YX, Jia YP. [Study of clinical outcome and prognosis in pediatric core binding factor-acute myeloid leukemia]. Zhonghua Xue Ye Xue Za Zhi. 2019 Jan 14;40(1):52-57. doi: 10.3760/cma.j.issn.0253-2727.2019.01.010. Chinese. PMID 30704229
- [Background] Minor EA, Kupec JT, Nickerson AJ, Narayanan K, Rajendran VM. Increased DMT1 and FPN1 expression with enhanced iron absorption in ulcerative colitis human colon. Am J Physiol Cell Physiol. 2020 Feb 1;318(2):C263-C271. doi: 10.1152/ajpcell.00128.2019. Epub 2019 Nov 13. PMID 31721611
- [Background] Peng Z, Xiang J, He Z, Zhang T, Xu L, Cui B, Li P, Huang G, Ji G, Nie Y, Wu K, Fan D, Zhang F. Colonic transendoscopic enteral tubing: A novel way of transplanting fecal microbiota. Endosc Int Open. 2016 Jun;4(6):E610-3. doi: 10.1055/s-0042-105205. Epub 2016 Apr 28. PMID 27556065
- [Background] Lu G, Wang W, Li P, Wen Q, Cui B, Zhang F. Washed preparation of faecal microbiota changes the transplantation related safety, quantitative method and delivery. Microb Biotechnol. 2022 Sep;15(9):2439-2449. doi: 10.1111/1751-7915.14074. Epub 2022 May 16. PMID 35576458